CLINICAL TRIAL: NCT03387189
Title: Morbidity of Second Stage Cesarean Sections Before and After Provider Completion of Simulation Education at Regions Hospital
Brief Title: Evaluation of a Quality Improvement Project on Impacted Fetal Head at Cesarean Section
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: Regions Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RG1700319
Record Dates: First submitted 2017-12-04; First posted 2018-01-02 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-01

CONDITIONS: Obstetric Labor Complications; Cesarean Section
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Quality Improvement Project (Pre-Period): Quality Improvement Project: Pre-Period (7/1/2016 to 12/31/2017) Patients received care at the intervention hospital in the 18 months before providers participated in the department-wide, simulation-based educational training.
- No Quality Improvement Project (Pre-Period): No Quality Improvement Project: Pre-Period (7/1/2016 to 12/31/2017) Patients received care at the comparison hospital where no quality improvement educational training had occurred.
- Quality Improvement Project (Post-Period): Quality Improvement Project: Post-Period (1/1/2018 to 6/30/2019) Patients received care at the intervention hospital in the 18 months after providers participated in the department-wide, simulation-based educational training.
  Interventions: Other: Quality Improvement Project
- No Quality Improvement Project (Post-Period): No Quality Improvement Project: Post-Period (1/1/2018 to 6/30/2019) Patients received care at the comparison hospital where no quality improvement educational training had occurred.

INTERVENTIONS:
Other: Quality Improvement Project — Simulation education conducted at Regions Hospital for a Quality Improvement project on delivery of impacted fetal head at cesarean section. This is a department-wide, simulation-based educational training required for all Regions Hospital Birth Center staff physicians, residents, nursing staff, and surgical techs.
  Groups: Quality Improvement Project (Post-Period)

SUMMARY:
This study is an evaluation of a Quality Improvement (QI) project addressing delivery of the impacted fetal head being conducted at Regions Hospital. This study aims to determine the morbidity of second stage cesarean deliveries before and after implementation of simulation protocols that address delivery of the impacted fetal head for Ob/gyn surgeons, nursing staff, and surgical technicians at Regions Hospital.

DETAILED DESCRIPTION:
Cesarean deliveries performed during the second stage of labor can be difficult due to impaction of the fetal head deep in the maternal pelvis and is associated with increased risk of both maternal and perinatal complications. There is little existing data to inform management of deeply impacted fetal heads, therefore these situations can be difficult for surgeons and other healthcare staff when they arise. Team simulations for obstetric emergencies have been shown to assist with provider comfort, improved clarity of thinking, and quicker action during emergency situations resulting in improved outcomes.

This study aims to show that a simulation education project for the entire obstetric team can decrease morbidity of difficult fetal head extraction associated with second stage cesarean deliveries and improve provider and nursing staff confidence regarding anticipation and management of this emergency. The simulation education project is not being conducted for the purpose of research, but is a department-wide educational activity and Quality Improvement project.

ELIGIBILITY:
Inclusion Criteria:

Patient: The patient study population includes all patients age 18-45 who underwent cesarean section during the second stage of labor (during the time period July 2016-June 2019 at Regions Hospital and Methodist Hospital) and their infants. Second stage is defined as the time between complete cervical dilation and delivery of the infant.

Medical staff: All staff members (staff physicians, residents, nurses, surgical technicians) at Regions Hospital who practice in the Birth Center who underwent required simulation education regarding delivery of impacted fetal heads during second stage cesarean section and completed the surveys as part of the QI project. Note: Medical staff were not enrolled in the research study; rather, staff survey data from the QI project was a data source for the study.

Exclusion Criteria:

Patient: Exclusion criteria include patients who underwent cesarean section in second stage for malpresentations (i.e., breech and noncephalic presentations) and patients who underwent cesarean section prior to 37 weeks gestation.

Medical staff: No exclusion criteria

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 1. Patients who underwent cesarean section during the second stage of labor and their infants.
  2. Medical staff who participated in the simulation-based educational training on impacted fetal head at cesarean section as part of the QI project.
     .
Sampling Method: Non-Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kamalini X Das, MD, Principal Investigator — HealthPartners Institute
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seal SL, Dey A, Barman SC, Kamilya G, Mukherji J, Onwude JL. Randomized controlled trial of elevation of the fetal head with a fetal pillow during cesarean delivery at full cervical dilatation. Int J Gynaecol Obstet. 2016 May;133(2):178-82. doi: 10.1016/j.ijgo.2015.09.019. Epub 2016 Jan 15. PMID 26868074
- [Background] Barrier BF, Allison JL, Andelin CO, Drobnis EZ. A simple device prevents hysterotomy extensions during cesarean delivery for failed second stage of labor. Gynecol Obstet Invest. 2013;76(2):90-4. doi: 10.1159/000351567. Epub 2013 May 24. PMID 23711893
- [Background] Jeve YB, Navti OB, Konje JC. Comparison of techniques used to deliver a deeply impacted fetal head at full dilation: a systematic review and meta-analysis. BJOG. 2016 Feb;123(3):337-45. doi: 10.1111/1471-0528.13593. Epub 2015 Aug 24. PMID 26301522
- [Background] Veisi F, Zangeneh M, Malekkhosravi S, Rezavand N. Comparison of "push" and "pull" methods for impacted fetal head extraction during cesarean delivery. Int J Gynaecol Obstet. 2012 Jul;118(1):4-6. doi: 10.1016/j.ijgo.2011.12.027. Epub 2012 Apr 27. PMID 22541809
- [Background] Berhan Y, Berhan A. A meta-analysis of reverse breech extraction to deliver a deeply impacted head during cesarean delivery. Int J Gynaecol Obstet. 2014 Feb;124(2):99-105. doi: 10.1016/j.ijgo.2013.08.014. Epub 2013 Nov 6. PMID 24290068

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Note: Medical staff were not enrolled in the research study; rather, staff survey data from the QI project was a data source for the study.
Pre-assignment Details: Study start date 1/1/2018, the first date in which a patient received care at the intervention hospital after staff received simulation training. The first 205 patients included in this study (7/1/2016-12/31/2017) were identified retrospectively and received care before the intervention. The next 204 patients (1/1/2018-6/30/2019) were included prospectively, post-implementation of the intervention. Only 73 of the 204 were exposed to providers that partook in the simulation.
Groups:
- Quality Improvement Project (Pre-Period): Simulation education conducted at Regions Hospital for a Quality Improvement project on delivery of impacted fetal head at cesarean section. This is a department-wide, simulation-based educational training required for all Regions Hospital Birth Center staff physicians, residents, nursing staff, and surgical techs. This arm includes patients who received care pre-period (7/1/2016 to 12/31/2017) who were cared for by providers who had yet to participate in the quality improvement project intervention.
- No Quality Improvement Project (Pre-Period): The comparison group is Methodist Hospital where the Quality Improvement project did not occur. This arm includes patients who received care pre-period (7/1/2016 to 12/31/2017). This group received care by providers who did not participate in the quality improvement project intervention.
- Quality Improvement Project (Post-Period): Quality Improvement Project: Simulation education conducted at Regions Hospital for a Quality Improvement project on delivery of impacted fetal head at cesarean section. This is a department-wide, simulation-based educational training required for all Regions Hospital Birth Center staff physicians, residents, nursing staff, and surgical techs. This arm includes patients who received care in the post-period (1/1/2018 to 3/20/2019) who were cared for by providers who had participated in the quality improvement project intervention.
- No Quality Improvement Project (Post-Period): No Quality Improvement Project: The comparison group is Methodist Hospital where the Quality Improvement project did not occur. This arm includes patients who received care post-period (1/1/2018 to 3/20/2019). This group received care by providers who did not participate in the quality improvement project intervention.
Period: Pre-Simulation (7/1/2016 to 12/31/2017)
Arm/Group | Quality Improvement Project (Pre-Period) | No Quality Improvement Project (Pre-Period) | Quality Improvement Project (Post-Period) | No Quality Improvement Project (Post-Period)
Started | 99 | 106 | 0 | 0
Completed | 99 | 106 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Post-Simulation (1/1/2018 to 6/30/2019)
Arm/Group | Quality Improvement Project (Pre-Period) | No Quality Improvement Project (Pre-Period) | Quality Improvement Project (Post-Period) | No Quality Improvement Project (Post-Period)
Started | 0 | 0 | 73 | 131
Completed | 0 | 0 | 73 | 131
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of second stage cesarean section procedures at each study site
Groups:
- Quality Improvement Project (Post-Period): Quality Improvement Project: Post-Period (1/1/2018 to 3/20/2019)
  Patients received care at the intervention hospital in the 18 months after providers participated in the department-wide, simulation-based educational training.
- No Quality Improvement Project (Post-Period): No Quality Improvement Project: Post-Period (1/1/2018 to 3/20/2019)
  Patients received care at the comparison hospital where no quality improvement educational training had occurred.
- Total: Total of all reporting groups
Arm/Group | Quality Improvement Project (Pre-Period) | No Quality Improvement Project (Pre-Period) | Quality Improvement Project (Post-Period) | No Quality Improvement Project (Post-Period) | Total
Number analyzed (Participants) | 99 | 106 | 73 | 131 | 409
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 99 | 106 | 73 | 131 | 409
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 106 | 73 | 131 | 409
  Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Maternal BMI [Mean (Standard Deviation); unit: kg/m^2] | 33.5 (5.9) | 33.5 (6.6) | 31.5 (6.7) | 32.7 (6.1) | 32.9 (6.3)
Fetal Weight [Mean (Standard Deviation); unit: grams] | 3619 (468) | 3609 (460) | 3534 (436) | 3526 (460) | 3571 (458)
Gestational Age at Time of C-Section [Mean (Standard Deviation); unit: Weeks] | 39.9 (1.2) | 40.3 (1) | 39.8 (1.3) | 40.1 (1.0) | 40.0 (1.1)
Length of Second Stage [Count of Participants; unit: Participants]
  0-2 hours | 20 | 17 | 11 | 20 | 68
  2-4 Hours | 37 | 32 | 22 | 46 | 137
  4+ Hours | 41 | 57 | 40 | 64 | 202
  Missing | 1 | 0 | 0 | 1 | 2
Cesarean Indication [Count of Participants; unit: Participants]
  Maternal | 73 | 81 | 44 | 90 | 288
  Fetal | 24 | 22 | 28 | 40 | 114
  Missing | 2 | 3 | 1 | 1 | 7
Previous C-Section (% yes) [Count of Participants; unit: Participants] | 17 | 10 | 7 | 21 | 55
Parity [Count of Participants; unit: Participants]
  0 | 72 | 87 | 54 | 105 | 318
  1 | 15 | 14 | 12 | 20 | 61
  2 | 9 | 5 | 0 | 5 | 19
  3 | 2 | 0 | 3 | 1 | 6
  4 | 0 | 0 | 3 | 0 | 3
  5+ | 1 | 0 | 1 | 0 | 2
Use of Tocolytics (% yes) [Count of Participants; unit: Participants] | 1 | 0 | 3 | 4 | 8
Type of Uterine Incision [Count of Participants; unit: Participants]
  Classical | 1 | 0 | 0 | 13 | 14
  Upper Lower Uterine Segment | 1 | 0 | 2 | 89 | 92
  Lower Lower Uterine Segment | 97 | 106 | 70 | 29 | 302
  Vertical Lower Uterine Segment | 0 | 0 | 1 | 0 | 1
Fetal Station [Count of Participants; unit: Participants] — Fetal station indicates how far the baby's head has descended into the pelvis in labor. The farther the baby's head has descended, indicated by higher values, the closer to delivery. Fetal station was assessed by pelvic exam. A value of 0 indicates that the baby's head was at the level of the ischial spine while negative values reflect the distance in centimeters above the ischial spine, and positive values distance below the ischial spine. This measure is purely descriptive and reflect specifics of the 2nd-stage procedure
  Participants
    -2 to -1 | 7 | 11 | 6 | 13 | 37
    0 to +1 | 64 | 57 | 50 | 89 | 260
    +2 to +3 | 27 | 37 | 17 | 29 | 110
    Missing | 1 | 1 | 0 | 0 | 2
Delivery Method [Count of Participants; unit: Participants]
  Standard | 77 | 96 | 63 | 117 | 353
  Push | 20 | 9 | 8 | 13 | 50
  Pull | 2 | 1 | 2 | 1 | 6
Use of Instrumentation [Count of Participants; unit: Participants]
  None | 92 | 88 | 68 | 118 | 366
  Tool (Vacuum or Forceps) | 7 | 17 | 4 | 13 | 41
  Missing | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Composite Variable of Maternal Morbidity of Second Stage Cesarean Section
Description: For each eligible procedure during the study timeframe, data retrospective programmatic and manual chart reviews was used to flag the presence of any of the following events:
  a) extension of uterine incision (yes/no), b) operative blood loss >1000 mL (yes/no), c) requirement of any blood transfusion during cesarean section (yes/no), d) wound infection within 6 weeks of cesarean section (yes/no), e) endometritis within 6 weeks of cesarean section (yes/no).
  These individual endpoints were used to compose a composite variable reflecting maternal morbidity associated with each second stage cesarean section procedure (unit of analysis). The primary outcome variable was coded as "1" if any of the above events were recorded (Yes, maternal morbidity/complication occurred) or "0" if none.
Time Frame: During the procedure through 6 weeks following the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Quality Improvement Project (Pre-Period) | Quality Improvement Project (Post-Period) | No Quality Improvement Project (Pre-Period) | No Quality Improvement Project (Post-Period)
Number analyzed (Participants) | 99 | 73 | 106 | 131
Participants | 64 | 39 | 38 | 59
Statistical Analysis 1: Comparison: Quality Improvement Project (Pre-Period) vs Quality Improvement Project (Post-Period) vs No Quality Improvement Project (Pre-Period) vs No Quality Improvement Project (Post-Period); Test type: Superiority — Alpha - 0.05; p = 0.031, Regression, Logistic; Adjusted for length of second stage cesarean section, fetal station, delivery method, use of instrumentation , parity, and gestational age; Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.17 to 0.91] — Y = Intervention + Time + Intervention*Time + Covariates. Provided estimation parameter is the OR from the interaction term and can be interpreted as the differential change in odds of outcome from pre to post period associated with the intervention

2. Primary Outcome: Composite Variable of Infant Morbidity of Second Stage Cesarean Section
Description: For each eligible procedure during the study timeframe, data retrospective programmatic and manual chart reviews was used to flag the presence of any of the following events:
  a) 5 minute APGAR score <7 (yes/no), b) NICU admission (yes/no), c) umbilical cord arterial pH <7.1 ph units (yes/no), d) fetal injury of cesarean delivery during the second stage of labor (yes/no).
  These individual endpoints were used to compose a composite variable reflecting infant morbidity associated with each second stage cesarean section procedure (unit of analysis). The primary outcome variable was coded as "1" if any of the above events were recorded (Yes, infant morbidity/complication occurred) or "0" if none.
  **APGAR score is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth. A score of 7, 8, or 9 is normal and is a sign that the newborn is in good health.
Time Frame: During the procedure through 6 weeks following the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Quality Improvement Project (Pre-Period) | Quality Improvement Project (Post-Period) | No Quality Improvement Project (Pre-Period) | No Quality Improvement Project (Post-Period)
Number analyzed (Participants) | 99 | 73 | 106 | 131
Participants | 64 | 39 | 38 | 59
Statistical Analysis 1: Comparison: Quality Improvement Project (Pre-Period) vs Quality Improvement Project (Post-Period) vs No Quality Improvement Project (Pre-Period) vs No Quality Improvement Project (Post-Period); Test type: Superiority — Alpha - 0.05; p = 0.465, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.53 to 4.03] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Operative Time
Description: Operative Time measured in minutes defined as skin incision to delivery - Only compared between time periods at Intervention hospital that received quality improvement educational training.
Time Frame: During the procedure
Population: As was pre-specified in the Study Protocol, only the participants who received care at the intervention hospital were assessed for this measure.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Quality Improvement Project (Pre-Period) | Quality Improvement Project (Post-Period)
Number analyzed (Participants) | 99 | 73
Minutes | 74.6 (33) | 63.2 (22)
Statistical Analysis 1: Comparison: Quality Improvement Project (Pre-Period); Test type: Superiority — alpha - 0.05; p = 0.01, t-test, 2 sided; Mean Difference (Final Values) = -11.4, 95% CI 2-sided [-20.4 to -2.5]

4. Secondary Outcome: Length of Stay
Description: Length of Stay for delivery - Only compared between time periods at Intervention hospital that received quality improvement educational training.
Time Frame: During the procedure through 6 weeks following the procedure
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Quality Improvement Project (Pre-Period) | Quality Improvement Project (Post-Period)
Number analyzed (Participants) | 99 | 73
Hours | 76.1 (23) | 75.1 (19)
Statistical Analysis 1: Comparison: Quality Improvement Project (Pre-Period) vs Quality Improvement Project (Post-Period); Test type: Superiority — Alpha - 0.05; p = 0.75, t-test, 2 sided; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-76.0 to 5.5]

5. Secondary Outcome: Time From Uterine Incision to Delivery
Description: Time from Uterine Incision to Delivery measured in minutes - Only compared between time periods at Intervention hospital that received quality improvement educational training.
Time Frame: During the procedure
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Quality Improvement Project (Pre-Period) | Quality Improvement Project (Post-Period)
Number analyzed (Participants) | 99 | 73
Minutes | 1.7 (2) | 1.2 (1)
Statistical Analysis 1: Comparison: Quality Improvement Project (Pre-Period) vs Quality Improvement Project (Post-Period); Test type: Superiority — Alpha - 0.05; p = 0.02, t-test, 2 sided; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.0 to -0.1]

6. Secondary Outcome: UTI During Maternal Admission
Description: UTI during Maternal Admission (% yes) - Only compared between time periods at Intervention hospital that received quality improvement educational training.
Time Frame: During the procedure through 6 weeks following the procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Quality Improvement Project (Pre-Period) | Quality Improvement Project (Post-Period)
Number analyzed (Participants) | 99 | 73
Participants | 0 | 0

7. Secondary Outcome: Urethral Injury
Description: Urethral Injury (% yes) - Only compared between time periods at Intervention hospital that received quality improvement educational training.
Time Frame: During the procedure through 6 weeks following the procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Quality Improvement Project (Pre-Period) | Quality Improvement Project (Post-Period)
Number analyzed (Participants) | 99 | 73
Participants | 0 | 1

8. Secondary Outcome: APGAR Score at 1 Minute
Description: APGAR score at 1 minute < 7 (% yes) - Only compared between time periods at Intervention hospital that received quality improvement educational training.
  **APGAR score is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth. A score of 7, 8, or 9 is normal and is a sign that the newborn is in good health.
Time Frame: During the procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Quality Improvement Project (Pre-Period) | Quality Improvement Project (Post-Period)
Number analyzed (Participants) | 99 | 73
Participants | 17 | 21
Statistical Analysis 1: Comparison: Quality Improvement Project (Pre-Period) vs Quality Improvement Project (Post-Period); Test type: Superiority — Alpha - 0.05; p = 0.10, Fisher Exact; Risk Difference (RD) = 0.116, 95% CI 2-sided [-0.01 to 0.24]

9. Secondary Outcome: Fetal Death
Description: Fetal Death (% yes) - Only compared between time periods at Intervention hospital that received quality improvement educational training.
Time Frame: During the procedure through 6 weeks following the procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Quality Improvement Project (Pre-Period) | Quality Improvement Project (Post-Period)
Number analyzed (Participants) | 99 | 73
Participants | 0 | 0

10. Secondary Outcome: Fetal Hyperbilirubinemia
Description: Fetal Hyperbilirubinemia (% yes) - Only compared between time periods at Intervention hospital that received quality improvement educational training.
Time Frame: During the procedure through 6 weeks following the procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Quality Improvement Project (Pre-Period) | Quality Improvement Project (Post-Period)
Number analyzed (Participants) | 99 | 73
Participants | 27 | 22
Statistical Analysis 1: Comparison: Quality Improvement Project (Pre-Period) vs Quality Improvement Project (Post-Period); Test type: Superiority — Alpha - 0.05; p = 0.81, Fisher Exact; Risk Difference (RD) = 0.028, 95% CI 2-sided [-0.12 to 17.8]

11. Secondary Outcome: Head Pushed up From Below Prior to Cesarean Section
Description: Head pushed up from below (% yes) - Only compared between time periods at Intervention hospital that received quality improvement educational training.
Time Frame: During the procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Quality Improvement Project (Pre-Period) | Quality Improvement Project (Post-Period)
Number analyzed (Participants) | 99 | 73
Participants | 14 | 11
Statistical Analysis 1: Comparison: Quality Improvement Project (Pre-Period) vs Quality Improvement Project (Post-Period); Test type: Superiority — Alpha - 0.05; p = 1.0, Fisher Exact; Risk Ratio (RR) = 0.01, 95% CI 2-sided [-0.11 to 0.13]

12. Secondary Outcome: Provider and Nurse Confidence Associated With Participation in Quality Improvement Training for Second Stage Cesarean Procedures
Description: Response on Likert Scale -
  * Not at all confident
  * Slightly confident
  * Moderately confident
  * Very confident Reported as % who responded they were very or moderately confident on each item - Only assessed in providers at the Intervention hospital that received quality improvement educational training.
Time Frame: Surveys distributed directly before, directly after, and 6 months after simulation training.
Population: The number of participants analyzed reflects a different denominator than other outcomes. This outcome was measured in medical staff at the intervention hospital who participated in the simulation training. We collected survey responses at three timepoints - Directly before participating in the simulation training, directly after participating in the simulation training, and six-months after completing the simulation training. The count of participants reflects the number of survey respondents.
Measure: Count of Participants; unit: Participants
Groups:
- Quality Improvement Project (Pre-Period): Providers/Nurse participants who responded to survey immediately before simulation training in winter of 2017.
- Quality Improvement Project (Post-Period): Providers/Nurse participants who responded to survey immediately post simulation training in winter of 2017
- Quality Improvement Project (6-Months-Post): Providers/Nurse participants who responded to survey six-months post simulation training
Arm/Group | Quality Improvement Project (Pre-Period) | Quality Improvement Project (Post-Period) | Quality Improvement Project (6-Months-Post)
Number analyzed (Participants) | 110 | 112 | 72
Participants
  Anticipating difficult extraction? | 56 | 90 | 62
  Performing your role during extraction? | 43 | 80 | 55
  Understand your role during obstetric emergency? | 57 | 98 | 68
  Understand role of others during emergency? | 50 | 100 | 65

ADVERSE EVENTS:
Time Frame: During the procedure through 6 weeks following the procedure
Description: Fetal death was collected as a secondary outcome for analysis. This will be reported as all-cause mortality. Serious and other AE were not defined as primary and secondary study outcomes describe any medical complication that occurred within sample.
Arm/Group | Quality Improvement Project (Pre-Period) | No Quality Improvement Project (Pre-Period) | Quality Improvement Project (Post-Period) | No Quality Improvement Project (Post-Period)
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/106 | 0/73 | 1/131
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/106 | 0/73 | 0/131
Other Adverse Events (participants affected / at risk) | 0/99 | 0/106 | 0/73 | 0/131

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT03387189/Prot_SAP_000.pdf